CLINICAL TRIAL: NCT02797873
Title: Emotional and Non-emotional Regulation in Patients With Emotional Instability Personality Disorder (EIP) and Attention Deficit Hyperactivity Disorder (ADHD) Symptoms
Brief Title: Emotional and Non-emotional Regulation in Patients With Emotional Instability and ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Predrag Petrovic, MD, PhD, Associate Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/127-31/1_EI_ADHD
Record Dates: First submitted 2016-04-27; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Emotional Instability Personality Disorder (Borderline Personality Disorder); Attention Deficit Hyperactivity Disorder; Healthy Controls
MeSH Terms: conditions — Borderline Personality Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EIP (Experimental): Patients from the DBT unit suffering from symptoms of Emotional Instability (n=30), with different levels of ADHD symptoms as assessed by questionnaires Brown-ADD, ASRS and SDQ.
  Interventions:
  * fMRI - Stroop task
  * fMRI - MID task
  * Stop Signal task
  * Structural T1 MRI scan
  * Structural T2 MRI scan
  * DTI MRI scan
  * Resting state MRI scan
  * FEFA 2
  * SCID-II
  * SDQ
  * ASRS
  * AQ
  * TAS-20
  * Raven's SPM
  * Reading ability
  * Ishihara's tests for colour deficiency
  * Additional questionnaire
  * Brown-ADD
  * MFQ
  * STAI-T
  * BIS
  * DAWBA
  * STAI-S
  * Sleepiness rating x 6
  * Motivation rating x 6
  Interventions: Other: fMRI - Stroop task; Other: fMRI - MID task; Behavioral: Stop Signal Task; Other: SCID-II; Other: SDQ; Other: ASRS; Other: AQ; Other: TAS-20; Other: Raven's SPM; Other: Reading ability; Other: Ishihara's tests for colour deficiency; Other: Additional questionnaire; Other: Brown-ADD; Other: MFQ; Other: STAI-T; Other: BIS; Other: DAWBA; Other: STAI-S; Other: Sleepiness rating; Other: Motivation rating; Behavioral: FEFA2; Other: Structural T1 MRI scan; Other: Structural T2 MRI scan; Other: DTI MRI scan; Other: Resting state MRI scan
- Healthy controls (Experimental): Matched healthy controls (according to age, IQ and socio economic status) recruited from high schools in Stockholm area (n=30).
  Interventions:
  * fMRI - Stroop task
  * fMRI - MID task
  * Stop Signal task
  * Structural T1 MRI scan
  * Structural T2 MRI scan
  * DTI MRI scan
  * Resting state MRI scan
  * FEFA 2
  * SCID-II
  * SDQ
  * ASRS
  * AQ
  * TAS-20
  * Raven's SPM
  * Reading ability
  * Ishihara's tests for colour deficiency
  * Additional questionnaire
  * Brown-ADD
  * MFQ
  * STAI-T
  * BIS
  * DAWBA
  * STAI-S
  * Sleepiness rating x 6
  * Motivation rating x 6
  Interventions: Other: fMRI - Stroop task; Other: fMRI - MID task; Behavioral: Stop Signal Task; Other: SCID-II; Other: SDQ; Other: ASRS; Other: AQ; Other: TAS-20; Other: Raven's SPM; Other: Reading ability; Other: Ishihara's tests for colour deficiency; Other: Additional questionnaire; Other: Brown-ADD; Other: MFQ; Other: STAI-T; Other: BIS; Other: DAWBA; Other: STAI-S; Other: Sleepiness rating; Other: Motivation rating; Behavioral: FEFA2; Other: Structural T1 MRI scan; Other: Structural T2 MRI scan; Other: DTI MRI scan; Other: Resting state MRI scan

INTERVENTIONS:
Other: fMRI - Stroop task — 2 x 10 minutes Stroop task (2 x 5 minutes emotional blocks, 2 x 5 minutes non-emotional blocks, order balanced across participants) performed during fMRI scan. See Detailed Study Description.
Other: fMRI - MID task — 2 x 10 minutes MID task performed during fMRI scan. See Detailed Study Description.
Behavioral: Stop Signal Task — Performed at a computer at first visit, 10 minutes divided into 3 blocks. See Detailed Study Description.
Other: SCID-II — See Detailed Study Description.
Other: SDQ — See Detailed Study Description.
Other: ASRS — See Detailed Study Description.
Other: AQ — See Detailed Study Description.
Other: TAS-20 — See Detailed Study Description.
Other: Raven's SPM — See Detailed Study Description.
Other: Reading ability — See Detailed Study Description.
Other: Ishihara's tests for colour deficiency — See Detailed Study Description.
Other: Additional questionnaire — including questions about somatic disease, current medication, BMI, smoking habits, first menstruation, last menstruation's first day, days without active oral contraceptive pill during last month, claustrophobia, vision impairment.
Other: Brown-ADD — See Detailed Study Description.
Other: MFQ — See Detailed Study Description.
Other: STAI-T — See Detailed Study Description.
Other: BIS — See Detailed Study Description.
Other: DAWBA — See Detailed Study Description.
Other: STAI-S — See Detailed Study Description.
Other: Sleepiness rating — Acquired 6 times while in MRI-scanner. See Detailed Study Description.
Other: Motivation rating — Acquired 6 times while in MRI-scanner. See Detailed Study Description.
Behavioral: FEFA2 — Assessing ability to recognise emotional face, performed at a computer at first visit. See Detailed Study Description.
Other: Structural T1 MRI scan — See Detailed Study Description and Outcome Measures.
Other: Structural T2 MRI scan — See Detailed Study Description.
Other: DTI MRI scan — See Detailed Study Description and Outcome Measures.
Other: Resting state MRI scan — See Detailed Study Description and Outcome Measures.

SUMMARY:
The purpose of this study is to investigate how emotional and non-emotional regulation processes differ in EIP patients (with different levels of ADHD symptoms/ADHD-comorbidity) compared to controls. The investigators will test these participants' abilities to regulate emotional and non-emotional processes, reward anticipation and reward receipt while they undergo functional magnetic resonance imaging (fMRI). The participants' motor inhibition capacity on a behavioral level will also be investigated.

The hypothesis is that EIP patients will present with more deficits in emotion regulation processes compared to controls, even when controlling for ADHD symptoms. It is also hypothesized that higher levels of ADHD symptoms will correlate with dysfunctional non-emotional regulation processes, on a behavioral as well as brain mechanistic level.

DETAILED DESCRIPTION:
Background: Comorbidity of Emotional Instability Personality Disorder (EIP) and Attention Deficit Hyperactivity Disorder (ADHD) is common, and the two patient groups partially exhibit similar problems. The main hypothesis is that the two disorders are mechanistically related. The investigators believe that the mechanisms underlying the problems are linked to two parallel regulating systems in the brain. Here, prefrontal and anterior cingulate systems are in focus. The first system - including the dorsolateral prefrontal cortex (dlPFC) and the caudal anterior cingulate cortex (cACC) - regulates non-emotional (and exteroceptive) information. The other system - including the lateral orbitofrontal prefrontal cortex (lObfc) and rostral anterior cingulate cortex (rACC) - regulates emotional (and interoceptive) information. The hypothesis is that the non-emotional/exteroceptive regulatory system is more affected in ADHD, while the emotional/interoceptive regulatory system is more affected in EIP.

Aims: The aim of this study is to differentiate between dysfunctional emotional regulation processes related to emotional instability symptoms (when controlling for non-emotional ADHD-like symptoms), and dysfunctional non-emotional regulation processes related to ADHD symptoms (when controlling for emotional instability symptoms).

Procedure:

* Participants: 30 young women from the Emotional Instability Unit at Child and Adolescent Psychiatry in Stockholm (Dialectic Behavioral Therapy unit ("DBT-teamet")), with traits of emotional instability and with varying levels of ADHD symptoms. 30 matched healthy controls.
* Tests:

Behavioral task: Stop Signal Task: measures participant's ability to inhibit a motor response. Outcome measures are Stop Signal Reaction Time (SSRT) and Go Reaction Time (GoRT)

fMRI task 1: Stroop task. Divided into 2 sessions of 10 minutes with 2 blocks in each. There are two types of blocks: Emotional Stroop task blocks (happy or fearful faces, with the word "HAPPY" or "FEAR" written across them) and Neutral Stroop task blocks (neutral faces of men and women with the word "MAN" or "WOMAN" written across them). Every other block is Emotional and every other is Neutral (balanced order between participants) so that each participant performs two emotional blocks and two neutral blocks. The task is to decide what emotion or gender is shown in the picture and ignore the word. Responses are made using a button box and reaction time is recorded for all the trials. Blood Oxygen Level Dependent (BOLD) signal is recorded in the brain during the task. Outcome measures are reaction times for the different trial types (incongruent(I) and congruent(C), also order dependent) as well as BOLD signal during these different types of trial.

fMRI task 2: Monetary Incentive Delay task (MID). Divided into 2 session of 10 minutes. Reward task in which the participant may win money (0 Swedish kronor (SEK), 10 SEK or 50 SEK in each trial). There is an anticipation phase in each trial, a response cue during which the participant needs to press a button as fast as she can, and an outcome phase in which feedback is presented of whether the participant has won the anticipated money or not. Outcome measures are BOLD activation during the anticipation phases of different levels of reward, and BOLD activation during the receipt/outcome phase of the different levels of reward. Reaction times for the different reward levels are also recorded.

The overall step-by-step procedure for each participant:

* Telephone screening (both participant and guardian): information about the study, MRI safety screening, check initial inclusion/exclusion criteria are met.
* Informed consent: sent by post to all legal guardians and the participant. Returned by post to test leader.
* The Strengths and Difficulties Questionnaire (SDQ) and socio-economic status questionnaires sent to one legal guardian and returned to test leader upon completion.
* Visit/Day 1: Assessment with questionnaires, interviews and behavioral testing (For selection of participants: Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV (SCID)-II interview Borderline and Antisocial parts, SDQ, Adult Self-Report Scale (ASRS), Autism Spectrum Quotient (AQ), Toronto Alexithymia Scale (TAS)-20, Ravens SPM, reading test, color vision test, questionnaire with additional questions. For characterization of participants: Brown-Attention Deficit Disorder (ADD), Mood and Feelings Questionnaire (MFQ), State and Trait Anxiety Inventory-Trait (STAI-T), Barratt's Impulsivity Scale (BIS)). Frankfurter Test und Training des Erkennens von fazialem Affekt (FEFA) 2 test (face recognition) and Stop signal test (SST). Approximately 3 hours.
* DAWBA computerized interview at home. Both participant and one legal guardian complete this.
* Additional information from patient records gathered, to verify current and previous diagnoses.
* Visit/Day 2: Assessments with questionnaires (STAI-S, last menstruation, sleepiness rating, motivation rating). MRI-scan: session 1: T1, Stroop session 1, Stroop session 2, T2. Break. Session 2: MID session 1, MID session 2. Break. Session 3: resting state, DTI. Assessments after scan: debriefing questionnaire, "After MID task" questionnaire. Approximately 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Undergone puberty
* Right-handed
* Monophasic contraceptives
* Speak Swedish fluently

Additional inclusion criteria EIP patients:

≥4/9 criteria of DSM-IV, measured by SCID-II interview

Exclusion Criteria:

* Impaired vision > +/- 5 D or other vision problem (squinting or severe astigmatism)
* BMI <17, BMI >35 due to possible hormonal disturbance
* Some medical drugs: benzodiazepines, neuroleptics, mood stabilisers, central stimulants, other neuro pharmaceuticals. (SSRIs are ok)
* Not suitable for MRI scan (metal implants or severe claustrophobia)
* AQ-score >26
* Alexithymia (≥52 in TAS20 questionnaire or poor score in facial recognition test (FEFA2));
* Mental retardation (IQ <70 according to Ravens SPM)
* Reading difficulties (reading speed >2 standard deviations slower than normal population of same age
* Established addiction problems (nicotine ok)
* Color blindness (>10 points on Ishihara-test)
* Psychotic disorder (according to medical history, DAWBA, medical records)
* Anorexia nervosa that has required hospital care
* Bipolar disorder (according to DAWBA and medical records)
* Neurological disease (according to medical history and medical records)
* Endocrinological disease
* Other disease, condition or treatment that may substantially affect cognition

Ages: 16 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
fMRI BOLD signal differences between groups - in Stroop task | Acquired during fMRI scan
  BOLD signal Neutral and Emotional blocks, and for Congruent and Incongruent trials (order dependent)
fMRI signal variations within patient group during Stroop task, depending on level of ADHD symptoms - in Stroop task | Acquired during fMRI scan
  BOLD signal Neutral and Emotional blocks, and for Congruent and Incongruent trials (order dependent)
Reaction times in Stroop task | Acquired during fMRI scan
fMRI BOLD signal differences between groups - in Monetary Incentive Delay task (MID) | Acquired during fMRI scan
  BOLD signal during anticipation phase of different levels of reward, and BOLD signal during receipt/outcome phase of different levels of reward.
fMRI BOLD signal differences within patient group during MID task, depending on level of ADHD symptoms - in MID task | Acquired during fMRI scan
  BOLD signal during anticipation phase of different levels of reward, and BOLD signal during receipt/outcome phase of different levels of reward.
Reaction times in MID task | Acquired during fMRI scan
Stop Signal reaction times (SSRT) from Stop Signal Task (SST) | Data necessary for estimation of SSRT acquired during fMRI scan

SECONDARY OUTCOMES:
Brown-ADD score | Acquired from questionnaire at first visit
Mood and Feelings questionnaire | Acquired from questionnaire at first visit
  dimensional measurement of depressive symptoms
STAI-T score | Acquired from questionnaire at first visit
  Measuring anxiety trait level
Barratt's impulsivity scale (BIS) | Acquired from questionnaire at first visit
STAI-S score | Baseline, acquired from questionnaire Day 2
  Measuring anxiety state level
Sleepiness score | Acquired during MRI scan, on Day 2
  Acquired 6 times in MRI scanner as follows: 1) Before first Stroop session. 2) Between Stroop session 1 and 2. 3) After Stroop session 2. 4) Before first MID session. 5) Between MID session 1 and 2. 6) After MID session 2.
Motivation score | Acquired during MRI scan, on Day 2
  Acquired 6 times in MRI scanner as follows: 1) Before first Stroop session. 2) Between Stroop session 1 and 2. 3) After Stroop session 2. 4) Before first MID session. 5) Between MID session 1 and 2. 6) After MID session 2.
Structural MRI data - volume | Acquired during MRI scan
Structural MRI data - surface area | Acquired during MRI scan
Structural MRI data - thickness | Acquired during MRI scan
Functional Connectivity (FC) | Acquired during resting state MRI scan
  Measuring the FC value between ROIs defined in hypothesis to determine strength of connectivity between these different brain regions.
Fractional Anisotropy (FA) of white matter | Acquired during Diffusion Tensor Imaging (DTI) scan

IPD SHARING:
Plan to Share IPD: Yes